CLINICAL TRIAL: NCT01185431
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Trial in Female Volunteers With Functional Constipation, to Evaluate the Improvement in Bowl Movement of Ficus Carica
Brief Title: The Effects of a Ficus Carica on Improvement in Bowl Movements in Female Volunteer With Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Study Director, Chae, Soo-wan, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTCF2_2010_YM
Record Dates: First submitted 2010-08-16; First posted 2010-08-20 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Functional Constipation
Keywords: Ficus Carica; Functional Constipation; Dietary Supplement; Fig Paste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ficus carica (Fig paste) (Experimental)
  Interventions: Dietary Supplement: Ficus carica (Fig paste)
- Control (Placebo paste) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (Placebo paste)

INTERVENTIONS:
Dietary Supplement: Ficus carica (Fig paste) — Ficus carica paste 300g/day
  Arms: Ficus carica (Fig paste)
Dietary Supplement: Placebo (Placebo paste) — Placebo composition 300g/day
  Arms: Control (Placebo paste)

SUMMARY:
This trial is being conducted to look for following changes when fig paste is taken by female subjects with functional constipation:

To evaluate the improvement of the bowel

To assess the quality of life and impact on female reproductive function

To evaluate the influence on glucose, cholesterol, HDL-cholesterol, LDL-cholesterol

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are female volunteers (unmarried), 19~40 years
* Subject who have functional constipation by ROME IIII criteria
* Subject who have over 36 hour colonic transit time
* Subject must provide written informed consent to participate in the study

Exclusion Criteria:

* Subject with a history or evidence of clinically significant gastrointestinal, anorectal, hepatic, renal, neurological, pulmonary, endocrine, blood tumor, psychiatric, Cardiovascular disease
* Subjects who have a gastrointestinal (GI) disease (Crohn's disease, etc.) that would increase the influence with absorbance medication or a GI surgery excluding appendectomy and hernia surgery
* Subject with uterine fibroids at ultrasonography
* Subject is pregnant, planning to become pregnant, or breast-feeding
* Subjects with childbearing potential (i.e. pre-menopausal, not surgically sterile) not willing to use a medically accepted contraceptive (oral contraception) regimen
* Known history of moderate to severe hepatic impairment (i.e., serum ALT>1.5×ULN, AST>1.5×ULN)
* Subjects with uncontrolled hypotension (indicated by a sitting systolic blood pressure ≤ 95 mmHg or diastolic blood pressure ≤ 60 mmHg measured) and hypertension (indicated by a sitting systolic blood pressure≥ 150 mmHg or diastolic blood pressure≥ 95 mmHg measured) at vital sign measurement
* Subjects with significant hypersensitivity about Ficus carica
* Subjects who received certain medications that cause the alteration of bowel movement within the past 2weeks prior to first administration
* Subjects who participated in other clinical investigation within 2 months prior to first administration
* Subject who drink constantly (21 units/week over)
* Subject who have Irritable bowel syndrome by ROME IIII criteria
* Any significant condition that, in the opinion of the investigator, could interfere with the subject's participation or compliance in the study (i.e., laboratory test and others)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Colonic transit time | 116 day
  Colonic transit time is measured in study visit 1 (as screening test), 3 (60day) and 5 (116day).

SECONDARY OUTCOMES:
Questionnaire for evacuation | 116 day
  Questionnaire include evacuation pattern (defecation frequency, times, senssation, abdominal displeasure, pain, stool shape, color)
Questionnaire for quality of life | 116 day
  Questionnaire include quality of life (physical function, limited role, pain, general healthy)
Questionnaire for woman reproductive function | 116 day
  Questionnaire include woman reproductive function (menstrual cycle, premenstrual syndrome)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea